CLINICAL TRIAL: NCT03153332
Title: Value of 3D Printing for Comprehension of Liver Surgical Anatomy
Status: Completed | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Collaborators: The Fifth People's Hospital of Dongguan City (Unknown); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Tianyou Yang, Principal Investigator, Guangzhou Women and Children's Medical Center
Other Study IDs: 3D printing
Record Dates: First submitted 2017-05-06; First posted 2017-05-15 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MDCT group: The MDCT images of seven hepatic tumors were loaded on software to uniform study conditions, allowing both axial and coronal scans visualization.
  Interventions: Other: surgical residents' comprehension of the hepatic anatomy
- 3D visualization system group: The 3D virtual reconstructions of seven hepatic tumors were loaded on the visualization software which enables the rotation of the virtual model.
  Interventions: Other: surgical residents' comprehension of the hepatic anatomy
- 3D printing group: 3D-printed models of seven hepatic tumors were created based on MDCT images, participants were allowed to freely handle them.
  Interventions: Other: surgical residents' comprehension of the hepatic anatomy

INTERVENTIONS:
Other: surgical residents' comprehension of the hepatic anatomy — Surgical residents were assigned to three different groups to evaluate different modes of patients' data. Residents were ask to state the liver segment in which the tumor resided and make a minimal resection proposal, including the tumor, the safety margin (1cm) and the dependent liver tissue. Residents were recommended to proceed in a classic way by resecting the whole liver segment. The time spent by each resident was also recorded in order to assess the quickness of comprehension and information transfer of the three different modes of presentation.

SUMMARY:
To our knowledge, it has not been analyze whether 3D printed liver model would improve the perception of a given liver tumor or the precision of operation planning in liver surgery. We design this prospective controlled trial to test whether the 3D-printed patient specific liver model could be more informative than standard MDCT (multi-row detector computed tomography ) and 3D visualization system in predicting the surgical anatomy of liver.

DETAILED DESCRIPTION:
The primary objective was to investigate whether 3D printing can improve localization of hepatic pathology. The secondary objective was to investigate whether 3D printing can improve the precision of surgical proposal.

The dataset of patients were prepared and stratified into MDCT, 3D visualization system and 3D printed liver model groups. The process started from MDCT scan image acquisition and moved through image segmentation and 3D rendering to end up with 3D printing.

Surgical residents were assigned to three different groups to study different modes of patients' data. Residents were ask to state the liver segment in which the tumor resides and make a minimal resection proposal, including the tumor, the safety margin (1cm) and the dependent liver tissue. Residents were recommended to proceed in a classic way by resecting the whole liver segment. The time spent by each resident was also recorded in order to assess the quickness of comprehension and information transfer of the three different modes of presentation.

ELIGIBILITY:
Inclusion Criteria:

* Surgical residents
* Must had experiences with MDCT and 3D visualization system

Exclusion Criteria:

* Non surgical residents
* No experiences with MDCT or 3D visualization system

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medical students had to finish five year medical school education (including one year internship), and then went into at least 3 year training program for surgical residency. Those who had finished training of general surgery were the study population.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
The primary outcomes was the precise allocation of hepatic disease | The primary outcome was assessed within 1 week after the collection of each participants' response.
  For tumor allocation to the liver segments, 8 points were awarded if all segments were correctly identified in which the tumors resided. If the tumors was located in more than one segment, the 8 maximal achievable points were divided between these segments. Erroneously identified segments were awarded 0 point. Alternatively, the primary outcomes were also simply judged as right or wrong according to the final surgical results.

SECONDARY OUTCOMES:
Resection proposal of liver pathology | The secondary outcome was assessed within 1 week after the collection of each participants' response.
  he resection proposals on the liver were compared with surgical results that had been evaluated by surgeons and judged by the formula mentioned earlier.
Time spent to judge tumor location | The secondary outcome was assessed within 1 week after the collection of each participants' response.
  The time spend to assess tumor location by each resident was documented as seconds

CONTACTS AND LOCATIONS:
Overall Officials: Tianyou Yang, MD, Principal Investigator — Guangzhou Women and Children's Medical Center, Guangzhou Medical University
Locations (1):
- he Fifth People's Hospital of Dongguan City, Dongguan, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Marescaux J, Clement JM, Tassetti V, Koehl C, Cotin S, Russier Y, Mutter D, Delingette H, Ayache N. Virtual reality applied to hepatic surgery simulation: the next revolution. Ann Surg. 1998 Nov;228(5):627-34. doi: 10.1097/00000658-199811000-00001. PMID 9833800
- [Result] Lamade W, Glombitza G, Fischer L, Chiu P, Cardenas CE Sr, Thorn M, Meinzer HP, Grenacher L, Bauer H, Lehnert T, Herfarth C. The impact of 3-dimensional reconstructions on operation planning in liver surgery. Arch Surg. 2000 Nov;135(11):1256-61. doi: 10.1001/archsurg.135.11.1256. PMID 11074877
- [Result] Zein NN, Hanouneh IA, Bishop PD, Samaan M, Eghtesad B, Quintini C, Miller C, Yerian L, Klatte R. Three-dimensional print of a liver for preoperative planning in living donor liver transplantation. Liver Transpl. 2013 Dec;19(12):1304-10. doi: 10.1002/lt.23729. Epub 2013 Oct 21. PMID 23959637
- [Result] Igami T, Nakamura Y, Hirose T, Ebata T, Yokoyama Y, Sugawara G, Mizuno T, Mori K, Nagino M. Application of a three-dimensional print of a liver in hepatectomy for small tumors invisible by intraoperative ultrasonography: preliminary experience. World J Surg. 2014 Dec;38(12):3163-6. doi: 10.1007/s00268-014-2740-7. PMID 25145821
- [Result] Kusaka M, Sugimoto M, Fukami N, Sasaki H, Takenaka M, Anraku T, Ito T, Kenmochi T, Shiroki R, Hoshinaga K. Initial experience with a tailor-made simulation and navigation program using a 3-D printer model of kidney transplantation surgery. Transplant Proc. 2015 Apr;47(3):596-9. doi: 10.1016/j.transproceed.2014.12.045. PMID 25891694
- [Result] Marconi S, Pugliese L, Botti M, Peri A, Cavazzi E, Latteri S, Auricchio F, Pietrabissa A. Value of 3D printing for the comprehension of surgical anatomy. Surg Endosc. 2017 Oct;31(10):4102-4110. doi: 10.1007/s00464-017-5457-5. Epub 2017 Mar 9. PMID 28281114